CLINICAL TRIAL: NCT04517656
Title: Biomarkers Impact Evaluation on the Post-transplant Immune Response After Allografting of Hematopoietic Stem Cells: MENTALO Study
Brief Title: Biomarkers Impact Evaluation on the Post-transplant Immune Response After Allografting of Hematopoietic Stem Cells
Acronym: MENTALO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other); Jean Monnet University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0601; 2020-A01901-38 (Other: N° IDRCB)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Malignant Hemopathy
Keywords: Allograft; Hematopoietic stem cells; Biomarkers; Immune response
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with hematologic malignancy (Experimental): Adult patient, over 18 years old, suffering from a malignant hemopathy (without exception) for whom an allogeneic hematopoietic stem cell transplant from a related or unrelated donor is indicated
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — A peripheral blood sample will be taken and will include 2 EDTA tubes of 5 mL, for a total volume of 10 mL:
  * Samples before the allograft,
  * Samples at different times post-allograft: 15 days, 30 days, 60 days, 90 days, 180 days, 360 days,
  * Samples in the event of the occurrence of concomitant events during the 12-month follow-up period: occurrence of acute Graft Versus Host Disease, chronic Graft Versus Host Disease, or relapse of the disease before the initiation of a new treatment.

SUMMARY:
Chemotherapy or targeted therapy are usually used to treat hematological pathologies. Despite of medical improvement, some of these pathologies present drug resistances, or high risk of relapse. Hematopoietic stem cell (HSC) transplantation remain the gold standard of consolidation, to maintain a durable response. In this situation, allograft with hematopoietic stem cells donor aims at producing Graft-versus-Tumor effect, by producing a new immune system, reproducing anti-tumoral immunity.

However, all hemopathies do not have the same sensibility. Nowadays, mechanisms underlying this phenomenon remain poorly understood.

Indeed, few data precisely document the expression of immunological checkpoints and other biomarkers in the context of allogeneic HSC transplantation, particularly their impact on post-transplant outcome.

DETAILED DESCRIPTION:
Chemotherapy or targeted therapy are usually used to treat hematological pathologies. Despite of medical improvement, some of these pathologies present drug resistances, or high risk of relapse. Hematopoietic stem cell (HSC) transplantation remain the gold standard of consolidation, to maintain a durable response. In this situation, allograft with hematopoietic stem cells donor aims at producing Graft-versus-Tumor effect, by producing a new immune system, reproducing anti-tumoral immunity.

However, all hemopathies do not have the same sensibility. Nowadays, mechanisms underlying this phenomenon remain poorly understood.

Indeed, few data precisely document the expression of immunological checkpoints and other biomarkers in the context of allogeneic HSC transplantation, particularly their impact on post-transplant outcome. Therefore, we want to systematically study the expression profile of different biomarkers during allogeneic transplantation, in order to establish a correlation between these expression patterns and post-transplant outcome. Ultimately, this research will enable to (i) have tools to predict the post-transplant response and (ii) define whether a targeted therapy could be beneficial or be contraindicated for adequate patient management.

Patients will be selected for the study once they meet all the inclusion criteria. The study will be proposed to them during the pre-allogeneic consultation as part of their usual care. This study does not modify the treatment or the usual management of patients according to the current practice of pre- and post-transplant management. Clinically, it consists of building up a relevant biological collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, over 18 years of age, suffering from a malignant hemopathy (without exception),
* Patient for whom an allogeneic hematopoietic stem cell transplant from a related or unrelated donor is indicated,
* Signed informed consent,
* Patient covered by a social security scheme.

Exclusion Criteria:

* Allogeneic hematopoietic stem cell transplantation from cord blood or haplo-identical transplant,
* Allogeneic transplant with post-transplant cyclophosphamide treatment,
* Allograft with sequential conditioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Expression level of Programmed death-ligand (PD) plasmatic biomarkers | 12 months
  Expression level of Programmed death-ligand (PD) plasmatic biomarkers will be quantified
Expression level of ST2 (suppression of tumourigenicity 2) plasmatic biomarkers | 12 months
  Expression level of ST2 (suppression of tumourigenicity 2) plasmatic biomarkers will be quantified
Expression level of Reg3 (regenerating islet-derived 3-alpha) plasmatic biomarkers | 12 months
  Expression level of Reg3 (regenerating islet-derived 3-alpha) plasmatic biomarkers will be quantified
Expression level of Elafin plasmatic biomarkers | 12 months
  Expression level of Elafin plasmatic biomarkers will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Cornillon, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No